CLINICAL TRIAL: NCT03697824
Title: Open-Label Phase 1b/2a Clinical Trial to Assess the Safety, Tolerability and Antitumor Activity of Genetically Engineered NY-ESO-1 Specific (c259) T Cells (GSK3377794) in Combination With Anti-Cancer Agents Including Pembrolizumab in HLA-A2+ Participants With NY-ESO-1 and/or LAGE-1a Positive Relapsed and Refractory Synovial Sarcoma
Brief Title: Clinical Trial of Safety, Tolerability and Antitumor Activity of Genetically Engineered T Cells in Combination With Anti-Cancer Agents in Relapsed and Refractory Synovial Sarcoma Expressing New York Esophageal Antigen-1 (NY-ESO-1) and/or LAGE-1a
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal decision, study will be replaced with a larger monotherapy trial
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209147
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Neoplasms
Keywords: HLA-A2+; Synovial Sarcoma; pembrolizumab; NY-ESO-1; GSK3377794; LAGE-1a
MeSH Terms: conditions — Neoplasms; Sarcoma, Synovial | interventions — pembrolizumab; fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm treatment study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK3377794+pembrolizumab (Experimental): After screening, eligible subjects will enter a leukapheresis phase, followed by lymphodepletion phase where they will be administered fludarabine and cyclophosphamide. On Day 1, subjects will receive a single dose of GSK3377794 administered as an intravenous infusion of 1 to 6 x10^9 total transduced cells. On Day 22, subjects will be administered pembrolizumab at a dose of 200 milligrams (mg) once every 3 weeks for adults and 2 mg/kilogram (kg) (up to 200 mg) once every 3 weeks for children for up to 35 cycles (2 years) or until subsequent disease progression.
  Interventions: Drug: GSK3377794; Drug: Pembrolizumab; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: GSK3377794 — GSK3377794 is genetically engineered NY-ESO-1 Specific (c259) T cells.
Drug: Pembrolizumab — Pembrolizumab will be administered at a dose of 200 mg once every 3 weeks for adults and 2 mg/kg (up to 200 mg) once every 3 weeks for children.
Drug: Fludarabine — Fludarabine will be used as a lymphodepleting chemotherapy.
Drug: Cyclophosphamide — Cyclophosphamide will be used as a lymphodepleting chemotherapy.

SUMMARY:
Adoptive T-cell therapy is a therapeutic approach that aims to generate an anti-tumor T-cell immune response by infusing a cancer subjects own T-cells obtained by leukapheresis, engineered and expanded in-vitro to express a tumor specific T-cell receptor. NY-ESO-1 and LAGE-1a antigens are tumor-associated proteins that have been found in several tumor types, including synovial sarcoma. This is an open-label study to evaluate the safety and efficacy of GSK3377794 (genetically engineered NY-ESO-1 Specific [c259] T Cells), in combination with anticancer agents including pembrolizumab in subjects with NY-ESO-1 and/or LAGE-1a positive relapsed and refractory synovial sarcoma. The study will consist of a target expression screening to determine if subjects are human leukocyte antigen (HLA)-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive and if their tumors express NY-ESO-1 and/or LAGE-1a, followed by a leukapheresis screening phase of up to 42 days prior to leukapheresis. Eligible subjects will enter a leukapheresis phase followed by lymphodepletion phase with cyclophosphamide and fludarabine. During the treatment phase, subjects will be administered GSK3377794 on Day 1 followed by pembrolizumab infusion once every 3 weeks from Day 22 (or Week 7) for up to 2 years. There will be a long-term follow-up phase from the end of treatment phase and for up to 15 years from the date of GSK3377794 administration.

ELIGIBILITY:
Inclusion Criteria:

* Target Expression Screening Phase: Subject must be >=10 years of age at the time of signing the informed consent. Younger subjects may only be enrolled upon consultation with Sponsor.
* Pathologically or histologically confirmed advanced synovial sarcoma that is either metastatic or unresectable and is either currently being treated with or has completed at least one line of standard chemotherapy regimen or subject is intolerant to it. Subjects can also undergo leukapheresis prior to initiating first line or standard therapy.
* Radiologically detectable disease.
* Life expectancy >=3 months.
* In the investigator's opinion, the subject is suitable for leukapheresis and, subsequently, for GSK3377794 and pembrolizumab infusion.
* An archival biopsy or fresh biopsy (if collected as part of standard of care) of tumor tissue is required to perform antigen expression analysis.
* Male or female subjects will be included. Contraception requirements will apply at the time of leukapharesis and treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol. For subjects <18 years of age (or the legal minimum age in the relevant country) their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion in order to obtain verbal assent.
* Leukapheresis Phase: In addition to the criteria mentioned above, the following criteria must also apply.
* Subject's tumor has been reviewed by the GlaxoSmithKline (GSK)-designated laboratory and confirmed as meeting the pre-defined threshold for expression of NY-ESO-1 and/or, if tested, LAGE-1a, using archival or fresh (if taken as standard of care) biopsy.
* HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 by high resolution testing.
* Left ventricular ejection fraction >=40%, or Fractional Shortening >=28%.
* Performance status: ECOG of 0-1 or for subjects <=10 years of age, Lansky >60.
* Subject must have adequate organ function 7 days prior to leukapheresis.
* Male or female subjects will be included. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. a) Male subjects are eligible to participate if they agree to the following during the intervention period starting at the first dose of chemotherapy for at least 12 months after receiving the T-cell infusion, or 4 months after there is no evidence of persistence/ gene modified cells in the subject's blood, whichever is longer. Must use effective contraception for at least 4 months after the last dose of pembrolizumab if this time frame is longer than the duration of contraception required in the context of chemotherapy and gene modified cells.
* Refrain from donating sperm and either: Be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier: a) Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant (as a condom may break or leak). b) Agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person.
* A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: a) Is not a WOCBP. OR, b) Is a WOCBP who will agree to use a barrier method (male condom) and use a contraceptive method that is highly effective (with a failure rate of <1% per year), during the intervention period and for at least 12 months after receiving the T-cell infusion, or 4 months after there is no evidence of persistence/ gene modified cells in the subjects blood, whichever is longer. WOCBP must use effective contraception for at least 4 months after the last dose of pembrolizumab if this time frame is longer than the duration of contraception required in the context of chemotherapy and gene modified cells. WOCBP should also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. c) A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before any dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the subject must be excluded from participation if the serum pregnancy result is positive. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Lymphodepletion and Treatment Phase: In addition to the criteria mentioned above, the following criteria must also apply:
* Subject has been treated with at least one line of standard chemotherapy regimen and is intolerant of or not actively responding to this regimen (i.e. the subject should not be taken prematurely off their primary regimen if they are continuing to respond to it).
* Subject must be presenting with at least two lesions: one measurable per RECIST 1.1 and the other required for biopsy. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Central nervous system (CNS) metastases with low CNS disease burden are allowed on a case by case basis after risk-benefit evaluation in consultation with the Sponsor Medical Monitor (or designee) if: a) Asymptomatic; b) Clinically stable; c) No history of bleeding within CNS metastases; d) No lesions in the brain stem; e) No untreated leptomeningeal metastases; f) No spinal cord compression; g) Not requiring escalating anti-epileptic treatment; h) Not requiring treatment with steroids; i) If treated with focal radiotherapy (for example, gamma knife radiosurgery), there is at least a 2-week wash-out period; j) Not treated with whole brain radiotherapy within the prior 4 weeks.
* Lymphodepleting regimen initiation is allowed if: a) There is clinical and/or radiographic evidence of disease progression; b) If supportive therapy (chemotherapy or radiotherapy) was used, the wash-out periods have been fulfilled; c) Supportive radiotherapy has not affected >25% of bone marrow; d) Following intermediate standard of care line of therapy.
* Another line of standard of care therapy may be administered between leukapheresis and treatment if: a) Indicated based on risk/benefit assessment and/or local regulatory requirements and following agreement with Sponsor's Medical Monitor (or designee); b) Treatments, adverse events and other clinical observations are reported in this study database
* A biopsy (excisional, incisional, or core) of tumor tissue obtained following cessation of the last line of treatment for synovial sarcoma but prior to initiating lymphodepleting chemotherapy is mandatory (if it is not feasible to obtain a fresh biopsy, archival tumor tissue is required).

Exclusion Criteria:

* Target Expression Screening Phase: Prior malignancy other than synovial sarcoma: a) Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. b) Subjects with previous malignancies that have been definitively treated, and have been in remission may be enrolled upon consultation with sponsor Medical Monitor or designee.
* Previous treatment with genetically engineered NY-ESO-1 specific T cells.
* Previous NY-ESO-1 vaccine.
* Prior gene therapy using an integrating vector.
* Previous allogeneic hematopoietic stem cell transplant.
* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the Investigator would compromise the subject's ability to tolerate protocol therapy or significantly increase the risk of complications.
* Leukapheresis Phase: In addition, to the above criteria subjects are not eligible for leukapharesis if any of the following criteria apply:
* Has chronic, recurrent, or active autoimmune/immune-mediated disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Uncontrolled intercurrent illness including, but not limited to: a) Ongoing or active infection requiring systemic therapy; b) Clinically significant cardiac disease defined by congestive heart failure New York Heart Association (NYHA) Class >1; c) Uncontrolled clinically significant arrhythmia in last 6 months; d) Acute coronary syndrome (angina or myocardial infarction) in last 6 months; e) Severe aortic stenosis or symptomatic mitral stenosis; f) Inadequate pulmonary function with mechanical parameters <40% predicted (Forced expiratory volume in 1 second [FEV1], Forced vital capacity [FVC], Total lung capacity [TLC], Diffusing capacity of the lung for carbon monoxide [DLCO]); g) Interstitial lung disease (subjects with existing pneumonitis as a result of radiation are not excluded; however, subjects cannot be oxygen dependent); h) Any other illness that in the judgment of the Investigator would compromise the subjects ability to tolerate protocol therapy or significantly increase the risk of complications
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment).
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Corrected QT interval duration (QTc) >450 milliseconds (msec) or QTc >480 msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read.
* Subject has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, fludarabine, other agents used in the study (Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule).
* Has severe hypersensitivity (>=Grade 3) to pembrolizumab and/or any of its excipients.
* Pregnant or breastfeeding females (due to risk to fetus or newborn).
* Any prior treatment-related toxicities must be CTCAE (Version 4.03) <=Grade 1 at the time of initiating study intervention (except for non-clinically significant toxicities e.g., alopecia, vitiligo). Subjects with Grade 2 toxicities that are deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled on a case-by-case basis in agreement between the Investigator and Sponsor's Medical Monitor (or designee).
* Other standard of care lines of therapy are allowed only if guidelines and wash-out periods are followed.
* Investigational treatment within 30 days or 5 half-lives (whichever is shorter) prior to leukapheresis. Investigational vaccines (other than NY-ESO-1 vaccines that are not allowed) must follow the wash-out period. Exceptions to this rule must be evaluated by the Investigator in agreement with the Sponsor's Medical Monitor (or designee).
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention. Subjects with positive Hepatitis C antibody due to prior resolved disease are can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained.
* A positive test for HIV antibody.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
* Lymphodepletion and Treatment Phase: In addition to the criteria mentioned above, subjects are not eligible for lymphodepletion or treatment if any of the following criteria apply: Subject has received cytotoxic therapy within 2 weeks prior to lymphodepleting chemotherapy: a. Subjects must have recovered from all AEs due to previous therapies to <=Grade 1 or Baseline. Subjects with <=Grade 2 neuropathy are eligible. b. Systemic corticosteroids or any other immunosuppressive therapy within 2 weeks prior to lymphodepleting chemotherapy.
* Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed.
* Major surgery <=28 days of first dose of study intervention.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2022-07-18 (Estimated); Study Completion 2022-07-18 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment limiting toxicities (TLT) | Up to 2 years
  The following toxicities will be considered as TLTs: Any >=Grade 4 adverse event (AE) except for Grade 4 fever and chills and Grade 4 hypoalbuminemia or abnormal electrolytes that are responding to supplementation/correction; Grade 3 non-infectious pneumonitis; Any other Grade 3 AE (excluding pneumonitis), that does not improve to Grade 2 within 7 days after onset despite medical management and supportive care; Any AE that permanently prevents subject from dosing with pembrolizumab in this trial.
Number of subjects with AEs | Up to 2 years
  An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Severity of AEs | Up to 2 years
  The severity of AEs will be graded according to National Cancer Institute-Common terminology criteria for adverse events (NCI-CTCAE) version 4.03.

SECONDARY OUTCOMES:
Number of subjects with serious adverse events (SAEs) | Up to 2 years
  An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; and other important medical events that may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Number of subjects with AE /SAEs leading to pembrolizumab administration delay, interruptions, and withdrawals | Up to 2 years
  Number of subjects with AE /SAEs leading to pembrolizumab administration delay, interruptions, and withdrawals will be summarized.
Number of subjects with abnormal hematology parameters | Up to 2 years
  Blood samples will be collected for the assessment of the following hematology parameters: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), reticulocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Number of subjects with abnormal clinical chemistry parameters | Up to 2 years
  Blood samples will be collected for the assessment of the following clinical chemistry parameters: blood urea nitrogen (BUN), creatinine, glucose, albumin, potassium, sodium, calcium, phosphorus, magnesium, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, lactate dehydrogenase (LDH), bicarbonate, total and direct bilirubin, total protein, chloride and urea.
Number of subjects with abnormal urine parameters | Up to 2 years
  Urine samples will be collected for the analysis of the following urine parameters: specific gravity, potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite and leukocyte esterase by dipstick.
Number of subjects with abnormal vital signs | Up to 2 years
  Vital signs will be measured in a semi-supine position after 5 minutes of rest and will include temperature, systolic and diastolic blood pressure, and pulse rate.
Eastern Cooperative Oncology Group (ECOG) performance scores | Up to 2 years
  For subjects >10 years of age, the performance status will be assessed using ECOG.
Lansky performance scores | Up to 2 years
  For subjects <=10 years of age, the performance status will be assessed using Lansky scale.
Number of subjects with abnormal electrocardiogram (ECG) parameters | Up to 2 years
  12-lead ECG will be obtained in triplicate using an automated ECG machine.
Overall Response Rate | Up to 2 years
  Overall response rate is defined as the percentage of subjects with a confirmed complete response (CR) or a partial response (PR) at any time as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression free survival | Up to 2 years
  Progression-free survival is defined as the time from the date of T-cell infusion until the earliest date of disease progression (PD) as assessed by the investigator per RECIST version 1.1, or death due to any cause.
Disease Control Rate | Up to 2 years
  Disease Control Rate is defined as the percentage of subjects with a confirmed CR, PR, or stable disease (SD) for at least 6 months as per RECIST version 1.1.
Duration of Response | Up to 2 years
  Duration of response is defined as the time from first documented evidence of CR or PR until the first documented sign of disease progression or death, in the subset of subjects who show a confirmed CR or PR.
Time to Response | Up to 2 years
  Time to response is defined as the time from the first dose to the first documented evidence of CR or PR for subjects with a confirmed CR or PR.
Maximum transgene persistence (Cmax) | Day -14 to Day -9, Days 1, 2, 4, 8, 15, 22, Weeks 5, 7 and once every 3 weeks from Week 10 to 106
  Peripheral blood samples will be collected at indicated time points for measurement of GSK3377794 transduced cell quantities. GSK3377794 T-cell persistence in the peripheral blood will be measured to establish the relationship between persistence and response to GSK3377794.
Time to Cmax (Tmax) | Day -14 to Day -9, Days 1, 2, 4, 8, 15, 22, Weeks 5, 7 and once every 3 weeks from Week 10 to 106
  Peripheral blood samples will be collected at indicated time points for measurement of GSK3377794 transduced cell quantities. GSK3377794 T-cell persistence in the peripheral blood will be measured to establish the relationship between persistence and response to GSK3377794.
Area under the time curve from zero to time t (AUC[0-t]) | Day -14 to Day -9, Days 1, 2, 4, 8, 15, 22, Weeks 5, 7 and once every 3 weeks from Week 10 to 106
  Peripheral blood samples will be collected at indicated time points for measurement of GSK3377794 transduced cell quantities. GSK3377794 T-cell persistence in the peripheral blood will be measured to establish the relationship between persistence and response to GSK3377794.
Number of subjects with NY-ESO-1/LAGE-1a expression in tumor tissues | Up to 2 years
  Biopsy of tumor tissue will be obtained to assess the tissue expression of the target antigen NY-ESO-1 and/or LAGE-1a.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com